CLINICAL TRIAL: NCT00175474
Title: Minimally Invasive Total Knee Arthroplasty Versus a Standard Surgical Technique: a Single-blinded Single-centre Randomized Controlled Trial
Brief Title: Comparison of a Minimally Invasive Technique for Total Knee Replacement to a Standard Technique
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C05-0036
Record Dates: First submitted 2005-09-11; First posted 2005-09-15 (Estimated); Last update posted 2011-10-14 (Estimated); Status verified 2011-10

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: knee surgery

SUMMARY:
Comparison of a minimally invasive technique for total knee replacement to a standard technique

ELIGIBILITY:
Inclusion Criteria:

* No inflammatory arthritis,
* no other lower limb problem,
* no major comorbidity

Exclusion Criteria:

-

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2005-09; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
length of stay

SECONDARY OUTCOMES:
Quality of life at 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bassam Masri, MD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada